CLINICAL TRIAL: NCT04419077
Title: Interest of Virtual Reality to Prevent Cancer Patient Anxiety Before Chemotherapy or an Invasive Act
Acronym: REV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL19_0992
Record Dates: First submitted 2020-03-02; First posted 2020-06-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Anxiety; Chemotherapy Effect; Breast Cancer; Head Cancer Neck
Keywords: Hypnosis
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Head and Neck Neoplasms | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Masking Description: 44 patients for the cohort " chemotherapy " and 22 patients for the cohort " invasive act ".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality exposure (Other): Virtual reality exposure just before an oncological procedure (invasive act or a chemotherapy)
  Interventions: Behavioral: Virtual reality exposure

INTERVENTIONS:
Behavioral: Virtual reality exposure — Patients will be exposed to a 10-20 min virtual reality session just before an oncological procedure (invasive act or chemotherapy).
  Patients will be able to choose between 4 virtual universes (beach, underwater, forest, space) and seven musical content.

SUMMARY:
The aim of the REV clinical trial is to evaluate the impact of a virtual reality exposure to decrease patient anxiety before chemotherapy or an invasive act. If positive, the access to virtual reality exposure is aimed to be used as standard of care at Lyon's hospital to improve cancer patient well-being in a drug-free manner.

The majority of cancer patients lives with high level of anxiety as soon as diagnosed. This level anxiety is particularly high before invasive acts but also before chemotherapy by side effects anticipation.

Hypnosis is a highly interesting drug-free approach to decrease patient's anxiety. It however requires on site specialists to be available whenever needed.

Virtual reality provides a distractive environment enabled to shift patient focus. It can support a switch of patient mindset by providing positive emotions.

Since 5 years, this disruptive technology is being more and more used as medical support thanks to a new generation of headsets enabling improved performance at cheaper prices.

Many publications have now demonstrated the positive impact of virtual reality to take in charge patients' pain or pre-operational anxiety.

DETAILED DESCRIPTION:
The primary objective of the REV study is to demonstrate the difference of anxiety before and after a virtual reality exposure using the State-Trait Anxiety Inventory (STAI-Y) before patients undergo an oncological procedure (invasive act or chemotherapy (C1D1).

The investigator's REV study aims to recruit 66 patients among three cohorts (22 patients per cohort) in 12 months.

* Breast cancer cohort (patient receiving an adjuvant or neoadjuvant chemotherapy with doxorubicin and cyclophosphamide)
* Head or neck cancer cohort (patient treated by concomitant radiochemotherapy)
* Cancer patient for which an invasive act inducing anxiety is planned (lumbar puncture, ascites puncture, thoracocentesis, myelogram, bone marrow biopsy, urinary catheterization, ..)

The REV study aims to impact Lyon's hospital patients' quality of life and well-being by decreasing their anxiety level during oncological treatments thanks to innovative supportive cares.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Patient Study Information and written informed consent
* Social Security Affiliation

For breast cancer cohort :

* Adult patient (>18 years)
* Histological or cytological proven breast cancer
* Eligible to an adjuvant or neo-adjuvant IV chemotherapy given every 2 to 3 weeks (with protocol doxorubicin- cyclophosphamide, docetaxel-cyclophosmadide, docetaxel-cyclophosphamide-trastuzumab, docetaxel, carboplatine, trastuzumab, epirubicin-cyclophosphamide, etc)
* Therapeutic strategy validated in multidisciplinary meeting
* First chemotherapy cure (C1D1) not initiated yet
* Patients with a complete healing after resection (for adjuvant chemotherapy)
* Patients that do not report residual pain with an intensity > 4.

For head, neck and bladder cancer cohort :

* Adult patient (>18 years)
* Histological or cytological proven head, neck or bladder cancer
* Patient eligible for an adjuvant or neoadjuvant based on cisplatin.
* Therapeutic strategy validated in multidisciplinary meeting
* First chemotherapy cure (C1D1) not initiated yet
* Patients with a complete healing after resection.
* Patients that do not report residual pain with an intensity > 4.

For invasive act leading to potential anxiety cohort :

* Adult patient (>18 years)
* Histological or cytological proven cancer
* Patient with a planned hospitalization at oncological unit
* Eupneic patient
* Afebrile patient

Patient for whom an invasive act leading to potential anxiety is planned (excluding percutaneous implantable chamber) :

* Puncture
* Deep biopsy
* Sounding
* Endoscopy without general anesthesia
* myelogram

Exclusion Criteria:

* Patient with a consciousness disturbance or a spatio-temporal disturbance
* Claustrophobic patient
* Patient with a non-stabilized psychiatric pathology
* Patient with seizure crisis background
* Patient with a visual or hearing disturbance that is not compatible with video watching and sound listening
* Patients with out-of range clinical parameters (arterial pressure, cardiac frequency,..)
* Patients with out-of range blood parameters that are not compatible with chemotherapy or an invasive act.
* Patient with a life expectancy below 3 months.
* Impossibility to track and follow patient (any reason)
* Patient deprived of liberty or subjected to guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Difference of anxiety using the State-Trait Anxiety Inventory before oncologic procedure | Before an invasive act or a chemotherapy
  Difference of anxiety before and after a virtual reality exposure using the State-Trait Anxiety Inventory (STAI-Y; A-State Scale) before patients undergo an oncologic procedure (invasive act or chemotherapy (C1D1).

SECONDARY OUTCOMES:
Difference of anxiety using a self-evaluation anxiety inventory before oncologic procedure | Before an invasive act or a chemotherapy
  Difference of anxiety before and after a virtual reality exposure using a self-evaluation anxiety inventory before patients undergo an oncologic procedure (invasive act or chemotherapy (C1D1).
  Comparison of responses between self-evaluation anxiety inventory before and after virtual reality exposure just before an oncologic procedure (invasive act or a chemotherapy)
Difference of anxiety using the State-Trait Anxiety Inventory before chemotherapy | Just before chemotherapy
  Difference of anxiety before and after a virtual reality exposure using the State-Trait Anxiety Inventory (STAI-Y; A-State Scale) or the Self-evaluation anxiety inventory before patients undergo chemotherapy (C1D1, C2D1, C3D1).
  Comparison of responses between the STAI-Y; A-State Scale or the Self-evaluation anxiety inventory before and after virtual reality exposure just before chemotherapy
Difference of anxiety using the State-Trait Anxiety Inventory before invasive act | Just before an invasive act
  Difference of anxiety before and after a virtual reality exposure using the State-Trait Anxiety Inventory (STAI-Y; A-State Scale) or the Self-evaluation anxiety inventory before patients undergo an invasive act.
  Comparison of responses between the STAI-Y; A-State Scale or the Self-evaluation anxiety inventory before and after virtual reality exposure just before an invasive act
Patient basal anxiety level just before an oncologic procedure | Just before an oncologic procedure
  Patient basal anxiety level using STAI-Y; A-State Scale, STAI-Y; Trait-State Scale or the Self-evaluation anxiety inventory just before an oncologic procedure (invasive act or a chemotherapy).
  Quotation of patient basal anxiety level using STAI-Y; A-State Scale, STAI-Y; Trait-State Scale or the Self-evaluation anxiety inventory just before an oncological procedure (invasive act or a chemotherapy)
Determination of patient anxiety level evolution through 3 cycles of chemotherapy | just before virtual reality exposure, after virtual reality exposure, after 1 hour of chemotherapy
  Determination of patient anxiety level evolution through 3 cycles of chemotherapy using the STAI-Y; A-State Scale and the Self-evaluation anxiety inventory (just before virtual reality exposure, after virtual reality exposure, after 1 hour of chemotherapy).
  Comparison of responses between the STAI-Y; A-State Scale and the Self-evaluation anxiety inventory before virtual reality exposure, after virtual reality exposure and after 1 hour of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'oncologie médicale, Institut de Cancérologie des Hospices Civils de Lyon, Hôpital Lyon sud, Pierre-Bénite, France